CLINICAL TRIAL: NCT03309423
Title: Utility of Mathematically Converted Venous to Arterial Blood Gas for Clinical Monitoring
Brief Title: Is Venous to Arterial Conversion (v-TAC) of Blood Gas Reliable in Critical Ill Patients in the ICU?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Mads Lumholdt, Principal investigator, Aalborg University
Other Study IDs: v-TAC-ICU
Record Dates: First submitted 2017-10-04; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Respiratory Insufficiency; Metabolic Disease; Acidosis; Alkalosis; Sepsis; Abdomen, Acute
Keywords: Blood gas analysis; Critical care; venus to arterial conversion
MeSH Terms: conditions — Respiratory Insufficiency; Metabolic Diseases; Acidosis; Alkalosis; Sepsis; Abdomen, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Respiratory disease: Patients with acute respiratory insufficiency admitted to the ICU and with pH <7,35 or >7,45
  Interventions: Diagnostic Test: venous to arterial conversion (v-TAC)
- Metabolic disease: Patients with acute metabolic disease admitted to the ICU and with pH <7,35 or >7,45
  Interventions: Diagnostic Test: venous to arterial conversion (v-TAC)
- Sepsis: Patients with acute sepsis admitted to the ICU and with pH <7,35 or >7,45
  Interventions: Diagnostic Test: venous to arterial conversion (v-TAC)

INTERVENTIONS:
Diagnostic Test: venous to arterial conversion (v-TAC) — Venous to arterial conversion (v-TAC) is a software (Obimedical, Denmark), which can convert venous blood gas values to arterial blood gas values. The principle of the method is a mathematical transformation of VBG values to arterialized values (aVBG) by simulating the transport of blood back through the tissue. To facilitate this simulation the following physiologically relevant assumptions were made: 1) The peripheral extremity was well perfused; 2) change in base excess across the tissue sampling site was approximately zero; 3) the respiratory quotient (rate of CO2 production and O2 utilisation over capillaries) could not vary outside the range 0.7 and 1.0, and 4) the haemoglobin concentration was constant from artery to vein.

SUMMARY:
Objective: Arterial blood gas (ABG) is essential in the clinical assessment of potential acutely ill patients venous to arterial conversion (v-TAC), a mathematical method, has recently been developed to convert peripheral venous blood gas (VBG) values to arterialized VBG (aVBG) values. The aim of this study is to test the reliability of aVBG compared to ABG in an intensive care unit (ICU) setting.

Method: Consecutive patients admitted to the ICU with pH values <7,35 or >7,45 are included in this study. Paired ABG and aVBG samples are drawn from patients via arterial catheter, central venous catheter and/or peripheral venous catheter and compared.

DETAILED DESCRIPTION:
Arterial blood gas (ABG) analysis is essential in assessment of respiratory and metabolic status in acutely ill patients. In comparison to peripheral venous blood (PVG) sampling, the ABG sampling procedure is more painful for the patient and technically more challenging for the clinician to perform. Other drawbacks of ABG sampling include adverse events such as subcutaneous hematoma, arterial thrombosis or embolization, and pseudoaneurysms.

Peripheral venous blood gas (VBG) sampling has been suggested as an alternative to the ABG procedure. This procedure causes less patient discomfort and the sample can be analysed in combination with other venous blood tests. Studies have revealed that pH and bicarbonate have good correlation, whereas venous and arterial blood gasses (pO2 and pCO2) show low agreement.

However, a new method has been developed to calculate ABG values mathematically from peripheral venous blood by use of venous to arterial conversion (v-TAC) software (Obimedical, Denmark), supplemented with oxygen saturation measured by pulse oximetry. The principle of the method is a mathematical transformation of VBG values to arterialized values (aVBG) by simulating the transport of blood back through the tissue. Initial testing of the method in an emergency department setting showed acceptable clinical congruence between arterial and mathematically arterialized pH and pCO2 with a small difference (+/- SD) on 0.001 +/- 0.024 and 0.00 0.46 kPa, respectively. However, inaccurate values of pO2 were seen when oxygen saturation measured by pulse oximetry was above 96%, due to the flat shape of the oxygen dissociation curve (ODC).

Although most patients in the ICU have arterial catheters therefrom ABG can be drawn, applying arterial catheter is difficult or even impossible in some patients. In relation to step-down some patients get arterial catheters removed and in the event of deterioration in patients acid-base or respiratory disease aVBG could prove useful as a minimally invasive tool to assess patients status.

The aim of this study is to investigate if v-TAC is reliable and safe to use in patients with critically respiratory or metabolic disease admitted to the ICU.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the intensive care with the following:
* Arterial catheter for other purpose.
* Peripheral venous catheter or central venous catheter for other purpose.

Exclusion Criteria:

* Normal pH in arterial blood gas.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to the ICU with acid-base and oxygenation parameters outside the normal reference values.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-01-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Lin's Concordance correlation coefficient (CCC) | 1. january 2018
  Comparison of pH between ABG and aVBG (from peripheral venous catheter). The closer CCC is to 1 the better correlation.
Lin's Concordance correlation coefficient (CCC) | 1. january 2018
  Comparison of pCO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from peripheral venous catheter). The closer CCC is to 1 the better correlation.
Lin's Concordance correlation coefficient (CCC) | 1. january 2018
  Comparison of pO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from peripheral venous catheter). The closer CCC is to 1 the better correlation.
Lin's Concordance correlation coefficient (CCC) | 1. january 2018
  Comparison of pH between ABG and aVBG (from central venous catheter). The closer CCC is to 1 the better correlation.
Lin's Concordance correlation coefficient (CCC) | 1. january 2018
  Comparison of pCO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from central venous catheter). The closer CCC is to 1 the better correlation.
Lin's Concordance correlation coefficient (CCC) | 1. january 2018
  Comparison of pO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from central venous catheter). The closer CCC is to 1 the better correlation.
Bland and Altman's plot | 1. january 2018
  Mean difference and 95% limits-of-agreement of pH between ABG and aVBG (from peripheral venous catheter)
Bland and Altman's plot | 1. january 2018
  Mean difference and 95% limits-of-agreement of pCO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from peripheral venous catheter).
Bland and Altman's plot | 1. january 2018
  Mean difference and 95% limits-of-agreement of pO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from peripheral venous catheter).
Bland and Altman's plot | 1. january 2018
  Mean difference and 95% limits-of-agreement of pH between ABG and aVBG (from central venous catheter).
Bland and Altman's plot | 1. january 2018
  Mean difference and 95% limits-of-agreement of pCO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from central venous catheter).
Bland and Altman's plot | 1. january 2018
  Mean difference and 95% limits-of-agreement of pO2 (Unit of Measurement: kilopascal) between ABG and aVBG (from central venous catheter).

SECONDARY OUTCOMES:
Number of patients with sepsis group. | 1. january 2018
  Number and percentage of patients in 'sepsis' group.
Number of patient with metabolic disease | 1. january 2018
  Number and percentage of patients in 'metabolic disease' group.
Number of patient with acute respiratory insufficiency | 1. january 2018
  Number and percentage of patients in 'respiratory disease group' group.
Mean number of days until pH neutrality in sepsis group | 1. january 2018
  Mean number of days until patients ABG pH was within the range 7.35-7.45 in 'sepsis' group.
Mean number of days until pH neutrality in patients with metabolic disease. | 1. january 2018
  Mean number of days until patients ABG pH was within the range 7.35-7.45 in 'metabolic disease' group.
Mean number of days until pH neutrality in patients with respiratory disease. | 1. january 2018
  Mean number of days until patients ABG pH was within the range 7.35-7.45 in 'respiratory disease' group.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Leutscher, Study Director — Professor, Center for Clinical Research
Locations (1):
- Faculty of Medicine, Doctoral School, Ph.d. study, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
IPD will be stored in safe government controlled data drives and paper data will be stored in a secure office. Doors to this office will be closed when investigators are not present. Sensitive IPD will not be shared with external researchers.